CLINICAL TRIAL: NCT01698385
Title: Prevention of Gestational Diabetes Through Lifestyle Modification (RADIEL) - a Randomized Controlled Multi-centre Intervention Study
Brief Title: Prevention of Gestational Diabetes Through Lifestyle Modification
Acronym: RADIEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); South Karelia, Social and Health Care District (Other)
Responsible Party: Principal Investigator, Saila Koivusalo, MD PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RADIEL
Record Dates: First submitted 2012-09-11; First posted 2012-10-03 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Active Comparator)
  Interventions: Other: Diet and exercise counseling
- Control, just measurements (No Intervention)

INTERVENTIONS:
Other: Diet and exercise counseling — diet and exercise counseling, setting of specific goals, follow-up of achievements, laboratory tests and measurements
  Other Names: Lifestyle intervention
  Arms: Lifestyle counseling

SUMMARY:
OVERALL OBJECTIVES:

1. To assess the efficacy of a diet and exercise intervention before and/or during pregnancy in the prevention of GDM and its fetal complications in women with high diabetes risk.
2. To assess the cost-effectiveness of a diet and exercise intervention in the prevention of GDM from a socio-economic point of view. To find out whether the intervention can be used to reduce health care costs due to GDM and T2DM.
3. To determine the long-term effectiveness of the above-mentioned lifestyle intervention in the reduction of T2DM incidence among women with prior GDM and their offspring

STUDY SUBJECTS Group 1: Women planning pregnancy with a history of diet/insulin-treated GDM or BMI >30 kg/m2. N= 250 + 250.

Group 2: Women in early pregnancy with a history of diet/insulin-treated GDM or BMI >30 kg/m2. N= 250 + 250

METHOD The Finnish multi-center randomized controlled intervention trial started in the maternity hospitals of Helsinki and Uusimaa District Area 1/2008 and in the South-Karelia Central Hospital in Lappeenranta in 9/2008. 1000 women at high GDM risk will be recruited. Half of the subjects are randomized into the intervention group and the other half act as controls receiving only standard antenatal care in addition to the laboratory tests taken and questionnaires administered by the RADIEL study.

The active intervention arm of the study will be carried out in a structured, standardized manner by diabetes nurses and nutritionists specifically trained for their tasks. The intervention includes:

1. Structured visits to diabetes nurse every 3 months before and during pregnancy as well as at 6 weeks, 6 and 12 months post partum. Visits include e.g. structured counseling on diet and exercise, setting of specific goals, follow-up of achievements, laboratory tests and measurements
2. Structured group visits to nutritionist at the moment of enrollment in the study, at the beginning of pregnancy as well as at 6 and 12 months post partum. Additional individual visits are booked if needed.
3. Services of physical activity advisors are provided by the study subjects' cities of residence free of charge to all who wish to receive extra counseling on exercise. If exercise goals are not met, study subjects book an appointment with the physical activity advisor.

LIFESTYLE TARGETS: 1.Weight: A weight loss of 5-10% before pregnancy if BMI > 25 and/or limited weight gain during the first two trimesters in pregnancy if BMI > 30. 2.Exercise: A minimum of 30 min. of exercise 5 times per week or 50 min. 3 times per week of moderate intensity exercise (Borg 11-15). Daily household and/or transportation physical activity. 3.Diet: Increased intake of vegetables, legumes, fruits and berries, whole grain and fiber, low-fat dairy, vegetable fats; and use of "plate model". Total energy intake: 1600-1800 kcal/day, with 40-50 E% carbohydrates, 30-40 E% fats, 20-25 E% protein.

MEASUREMENTS of maternal variables:

AT THE MOMENT OF ENROLMENT TO THE STUDY, and every 3 months before pregnancy:

(1) Waist circumference, blood pressure, pulse, weight, height (2) i.e. 2-hour OGTT, fP-insulin, fP-glucose, , GHbA1c, lipids, P-hCRP, P-IL-6, S-A1Glypr, leptin. (3) Background questionnaire (4) 15-D-questionnaire: health-related quality of life. (7) Food diary (2+1). Exercise diaries daily for one week.

PREGNANCY At the end of each trimester: (1) The same tests and measurements as in pre-pregnancy period. 2h-OGTT at H10-14 and at H24-28. (2) Questionnaire, 15-D questionnaire, EDPS (=Edinburgh post-partum depression scale) questionnaire for screening mood disorders at H10-13. (4) Food diaries (2+1), and exercise diaries daily for one week at H10-13 and H34-36.

POST PARTUM PERIOD (Groups 1-2) At 6 weeks, 6 and 12 months post partum: (1) The same follow-up tests and measurements as at the beginning. Lipids checked only at 12 months post partum. (2) 2-hour OGTT 6 weeks and 12 months post partum (3) Questionnaires at all visits. (5) Food and exercise diaries at 12 months post partum.

MEASUREMENTS of child's variables at birth

(1) weight (2) height (3) head circumference (4) From delivery records: Mode of delivery, Apgar scores, any perinatal complications, operations, need of neonatal intensive care and length of hospital. (3) Laboratory tests from cord blood.

TIMETABLE Recruitment started in February 2008 and ended in autumn 2011 when about 800 subjects had been recruited to the study. Intervention will continue until 2014 (including pre- and postpartum periods). Long-term follow up of both mothers' and children's cohorts starts in 2014 and has been planned to continue up to 10 years postpartum. Data analysis starts in autumn of 2013 and results will be reported from 2014 onwards in international peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI > 30)
* previous GDM

Exclusion Criteria:

* Age < 18 years
* diabetes before pregnancy
* medication influencing glucose homeostasis
* hypertension
* multiple pregnancy
* physical disability
* substance abuse
* severe psychiatric disorders
* significant co-operation difficulties

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2008-02; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in oral glucose tolerance test at variable time frames | 1) Baseline (group 1= planning a pregnancy; group 2=at gest.week 10-14); 2) at gest.week 10-14 (group 1) and 3) at gest.week 24-28; 4) 6 weeks and 12 months post partum

SECONDARY OUTCOMES:
Change from Baseline in weight at variable time frames | 1) Baseline (group 1= planning a pregnancy; group 2=at gest.week 10-14); 2) at gest.week 10-14 (group 1) and 3) at gest.week 24-28 and 34-36, and 4) 6 weeks, 6 months and 12 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Saila B Koivusalo, MD, Principal Investigator — University of Helsinki
Locations (1):
- Hospital District of Helsinki and Uusimaa, Helsinki, Finland

REFERENCES:
- [Derived] Blanco Sequeiros E, Tuomaala AK, Tabassum R, Bergman PH, Koivusalo SB, Huvinen E. Early ascending growth is associated with maternal lipoprotein profile during mid and late pregnancy and in cord blood. Int J Obes (Lond). 2023 Nov;47(11):1081-1087. doi: 10.1038/s41366-023-01361-x. Epub 2023 Aug 17. PMID 37592059
- [Derived] Huvinen E, Lahti J, Klemetti MM, Bergman PH, Raikkonen K, Orho-Melander M, Laivuori H, Koivusalo SB. Genetic risk of type 2 diabetes modifies the effects of a lifestyle intervention aimed at the prevention of gestational and postpartum diabetes. Diabetologia. 2022 Aug;65(8):1291-1301. doi: 10.1007/s00125-022-05712-7. Epub 2022 Apr 30. PMID 35501401
- [Derived] Huvinen E, Tuomaala AK, Bergman PH, Meinila J, Tammelin T, Kulmala J, Engberg E, Koivusalo SB. Ascending Growth is Associated with Offspring Adiposity in Pregnancies Complicated with Obesity or Gestational Diabetes. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e1993-e2004. doi: 10.1210/clinem/dgaa979. PMID 33524144
- [Derived] Huvinen E, Engberg E, Meinila J, Tammelin T, Kulmala J, Heinonen K, Bergman P, Stach-Lempinen B, Koivusalo S. Lifestyle and glycemic health 5 years postpartum in obese and non-obese high diabetes risk women. Acta Diabetol. 2020 Dec;57(12):1453-1462. doi: 10.1007/s00592-020-01553-1. Epub 2020 Jul 25. PMID 32712801
- [Derived] Valkama AJ, Meinila J, Koivusalo S, Lindstrom J, Rono K, Stach-Lempinen B, Kautiainen H, Eriksson JG. The effect of pre-pregnancy lifestyle counselling on food intakes and association between food intakes and gestational diabetes in high-risk women: results from a randomised controlled trial. J Hum Nutr Diet. 2018 Jun;31(3):301-305. doi: 10.1111/jhn.12547. Epub 2018 Feb 7. PMID 29468749
- [Derived] Huvinen E, Eriksson JG, Koivusalo SB, Grotenfelt N, Tiitinen A, Stach-Lempinen B, Rono K. Heterogeneity of gestational diabetes (GDM) and long-term risk of diabetes and metabolic syndrome: findings from the RADIEL study follow-up. Acta Diabetol. 2018 May;55(5):493-501. doi: 10.1007/s00592-018-1118-y. Epub 2018 Feb 19. PMID 29460080
- [Derived] Huvinen E, Koivusalo SB, Meinila J, Valkama A, Tiitinen A, Rono K, Stach-Lempinen B, Eriksson JG. Effects of a Lifestyle Intervention During Pregnancy and First Postpartum Year: Findings From the RADIEL Study. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1669-1677. doi: 10.1210/jc.2017-02477. PMID 29409025
- [Derived] Koivusalo SB, Rono K, Klemetti MM, Roine RP, Lindstrom J, Erkkola M, Kaaja RJ, Poyhonen-Alho M, Tiitinen A, Huvinen E, Andersson S, Laivuori H, Valkama A, Meinila J, Kautiainen H, Eriksson JG, Stach-Lempinen B. Gestational Diabetes Mellitus Can Be Prevented by Lifestyle Intervention: The Finnish Gestational Diabetes Prevention Study (RADIEL): A Randomized Controlled Trial. Diabetes Care. 2016 Jan;39(1):24-30. doi: 10.2337/dc15-0511. Epub 2015 Jul 29. PMID 26223239
- [Derived] Miettinen HE, Rono K, Koivusalo S, Stach-Lempinen B, Poyhonen-Alho M, Eriksson JG, Hiltunen TP, Gylling H. Elevated serum squalene and cholesterol synthesis markers in pregnant obese women with gestational diabetes mellitus. J Lipid Res. 2014 Dec;55(12):2644-54. doi: 10.1194/jlr.P049510. Epub 2014 Oct 9. PMID 25301963
- [Derived] Rono K, Stach-Lempinen B, Klemetti MM, Kaaja RJ, Poyhonen-Alho M, Eriksson JG, Koivusalo SB; RADIEL group. Prevention of gestational diabetes through lifestyle intervention: study design and methods of a Finnish randomized controlled multicenter trial (RADIEL). BMC Pregnancy Childbirth. 2014 Feb 14;14:70. doi: 10.1186/1471-2393-14-70. PMID 24524674